CLINICAL TRIAL: NCT06915948
Title: Postoperative Anatomical Closure of Idiopathic Chronic Giant Macular Hole on the Same Day Determined by Spectral Domain Optical Coherence Tomography for Macular Hole Surgery With Silicone Oil Tamponade
Brief Title: Postoperative Same Day Closure of Giant Macular Hole With Silicone Oil
Acronym: GiantMH-SO
Status: Completed | Type: Observational
Sponsor: Ahalia Foundation Eye Hospital (Other)
Responsible Party: Principal Investigator, Dr. Saurav Mahajan, Principal Investigator, Clinical Professor Adjunct, Ahalia Foundation Eye Hospital
Other Study IDs: 202103.; U1111-1312-4425 (Other: WHO UTN)
Record Dates: First submitted 2024-08-24; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Macular Holes; Vitrectomy
Keywords: Macular Hole; Giant Large Macular Hole; Silicone Oil; SD-OCT
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Macular Hole Surgery — Pars Plana Vitrectomy with ILM peeling with silicone oil tamponade

SUMMARY:
Patients with stage 3 and 4 macular holes of size >700 microns who underwent pars plana vitrectomy, Internal limiting Membrane peeling and silicone oil tamponade were followed at day 1 , 2 weeks and 1 month post silicone oil removal and anatomical closure of macular hole assessed at all intervals

DETAILED DESCRIPTION:
Patients who attended Retina OPD in Ahalia Foundation Eye Hospital, Palakkad were selected to participate in the study

Basic demographic profile which includes name, age, gender , address was noted .

Structured questionnaire was used to collect information about the presence of any systemic risk factors like diabetes mellitus, hypertension, any prior retinal surgery and high myopia .

Preoperatively , all subjects will be tested for BCVA , intraocular pressure measurement, slit lamp bio-microscopy of anterior segment and indirect non contact bio-microscopy of the fundus with 20D lens will be documented .

Using spectral domain optical coherence tomography diagnosis of macular hole was confirmed and hole form factor and diameter hole index calculated based on the findings in optical coherence tomography.

Patients with stage 3 and 4 macular holes of size >700 u who underwent pars plana vitrectomy, ILM peeling and silicone oil tamponade were shortlisted.

Patients follow up was done on day 1, 2 weeks and 1 month post silicone oil removal .

For each follow up , BCVA with silicon oil and intraocular pressure was measured and indirect noncontact bio-microscopy examination of the macula was examined. Assessment of macula was done using OCT on day 1, 2 weeks and 1 month post silicone oil removal .

In all patients the anatomical closure of macular hole was assessed on day 1, 2 weeks and 1 month post silicone oil removal .

Statistical methods

* The information recorded on the data collection forms were uploaded in an excel sheet and data were analyzed using IBM SPSS version 20.
* To obtain the characteristic of categorical variables, frequency and percentage were applied.
* To obtain the characteristic of numerical variables, mean and standard deviation were used.
* Chi square test/ Fisher's exact test was used to find association between HFF, DHI, gender with hole closure type of closure.
* Students t test and Man Whitney U test were performed to compare the average values of numerical parameters such as age, BCVA with hole closure, type of closure, HFF, DHI.
* Paired t test was used to compare the pre-Op and Final BCVA. P-value <0.05 was consideredto denote statistical significance.
* ANOVA was used wherever we had to compare numerical data/means between 3 groups of type of hole closure- open vs type I vs type II closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic chronic giant macular hole more than 700 micron size confirmed by indirect biomicroscopy and optical coherence tomography.
* Patients who give a valid informed consent
* Patients who underwent surgery

Exclusion Criteria:

* High myopic patients ( >10 D)
* Patients with history of ocular trauma
* Patients with history of any macular surgery
* Rhegmatogenous retinal detachment associated with macular hole
* Patients having vision loss due to other ocular comorbidities- glaucoma , macular pathology or vitreous hemorrhage.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -Patients (South Indians) who attended Retina OPD in Ahalia Foundation Eye Hospital, Palakkad, Kerala was selected to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of eyes with Immediate Anatomical Closure of Macular hole | Day 1
  Percentage (%) of eyes with Immediate Anatomical Closure of Macular hole on same day
Percentage of eyes having Type I Closure of Macular hole | Day 1; 2 weeks after surgery ; 1 month post silicone oil removal
  * Percentage (%) of eyes having Type I Closure of Macular hole at Day 0
  * Percentage (%) of eyes having Type I Closure of Macular hole at 2 weeks
  * Percentage (%) of eyes having Type I Closure of Macular hole 1 month post Silicone oil removal in eyes undergoing Silicone oil removal
Percentage of eyes having Type II Closure of Macular hole | At Day 1, 2 weeks after surgery and 1 month post Silicone oil removal
  * Percentage (%) of eyes having Type II Closure of Macular hole at Day 0
  * Percentage (%) of eyes having Type II Closure of Macular hole at 2 weeks
  * Percentage (%) of eyes having Type II Closure of Macular hole 1 month post Silicone oil removal in eyes undergoing Silicone oil removal
Percentage of eyes having Open Macular hole | At Day 1, 2 weeks after surgery and 1 month post Silicone oil removal
  * Percentage (%) of eyes having Open Macular hole at Day 0
  * Percentage (%) of eyes having Open Macular hole at 2 weeks
  * Percentage (%) of eyes having Open Macular hole 1 month post Silicone oil removal in eyes undergoing Silicone oil removal
Adverse events | Day 1
  Any adverse events

SECONDARY OUTCOMES:
Percentage of eyes with Anatomical Closure of Macular hole | 2 weeks post surgery , 1 month Post Silicone oil removal
  * Percentage (%) of eyes with Anatomical Closure of Macular hole at 2 week follow up
  * Percentage (%) of eyes with Anatomical Closure of Macular hole at 1 month post silicone oil removal
Role of Hole Forming Factor (HFF) in predicting Hole Closure | at day 1, 2 weeks post surgery
  * Number of eyes with HFF <0.5 achieving hole closure
  * Number of eyes with HFF >0.5 achieving hole closure
Role of Diameter Hole Index (DHI) in predicting Hole Closure | at day 1, 2 weeks post surgery
  * Number of eyes with DHI <0.5 achieving hole closure
  * Number of eyes with DHI >0.5 achieving hole closure
Mean Diameter Hole Index | 2 weeks post surgery
  * Mean Preoperative Diameter Hole Index(DHI) in eyes with Type I closure of macular hole
  * Mean Preoperative Diameter Hole Index(DHI) in eyes with Type II closure of macular hole
  * Mean Preoperative Diameter Hole Index(DHI) in eyes with Open macular hole
Mean Hole Forming Factor | 2 weeks post surgery
  * Mean Preoperative Hole Forming Factor(HFF) in eyes with Type I closure of macular hole
  * Mean Preoperative Hole Forming Factor(HFF) in eyes with Type II closure of macular hole
  * Mean Preoperative Hole Forming Factor(HFF) in eyes with Open macular hole
Visual Outcomes | Pre-operative (baseline) and 1 month post Silicone oil removal
  Visual Acuity In LogMAR (logarithm of the Minimum Angle of Resolution) units Pre-operatively (baseline) and after 1 month of silicone oil removal excluding eyes that needed resurgery
Resurgeries | 6 months
  No. of eyes that underwent resurgery for open macular hole No. of eyes that underwent resurgery for reason other than open macular hole
Reopened Holes | 6 months
  Number of hole reopen cases , even under silicone oil
Adverse events | 3 months
  Any adverse events in 3 months follow up .
Face down positioning | 1 month
  To find out relevance for maintaining face down positioning

CONTACTS AND LOCATIONS:
Overall Officials: Rajkumar Maheshwari, MS, Principal Investigator — Ahalia Foundation Eye Hospital; Amrutha S, DNB, Principal Investigator — Ahalia Foundation Eye Hospital; Saurav Mahajan, MS, Principal Investigator — Ahalia Foundation Eye Hospital; Sajeev C Jacob, MS, Study Chair — Ahalia Foundation Eye Hospital
Locations (1):
- Ahaliafoundation Eye Hospital, Palakkad, Kerala, India

IPD SHARING:
Plan to Share IPD: No